CLINICAL TRIAL: NCT00472303
Title: A Randomized Withdrawal, Active- and Placebo-controlled, Double-blind, Multi-center Phase III Trial Assessing Safety and Efficacy of Oral CG5503 (Tapentadol) PR* in Subjects With Moderate to Severe Chronic Malignant Tumor-related Pain
Brief Title: A Study to Evaluate Tapentadol (CG5503) in the Treatment of Chronic Tumor-Related Pain Compared With Placebo and Morphine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Grünenthal GmbH (Industry)
Collaborators: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 761101; 2006-004997-28 (EudraCT Number); KF5503/15 (Other: Grünenthal)
Record Dates: First submitted 2007-05-10; First posted 2007-05-11 (Estimated); Results first posted 2014-05-07 (Estimated); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Tumor; Pain
Keywords: Opioid; Central acting analgesic; CG5503 PR; Tumor related pain; Cancer related pain; Morphine; Pain assessment; Placebo
MeSH Terms: conditions — Neoplasms; Pain; Cancer Pain | interventions — Tapentadol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Matching Placebo after Tapentadol in Titration Phase (Placebo Comparator): Oral Tapentadol 100 mg to 250 mg twice daily. Participants randomized to placebo in the maintenance phase received 100 mg tapentadol prolonged release twice daily for 3 days to taper them off the tapentadol dose they had received in the Titration Phase. From the 4th day (Day 18) all participants received matching placebo in the maintenance (i.e. randomized withdrawal) phase.
  Interventions: Drug: Tapentadol Extended Release; Drug: Matching Placebo after Tapentadol in the Titration Phase.
- Morphine Controlled Release (Active Comparator): Oral Morphine 40 mg to 100 mg twice daily. Capsule taken orally, twice daily, morning & evening with preferably 12 hours (not less than 6 hours) between doses. Maintenance phase: continuing on dose level established in titration phase.
  Interventions: Drug: Morphine Sulphate Controlled Release
- Tapentadol Prolonged Release (Experimental): Oral Tapentadol 100 mg to 250 mg twice daily. Tablet taken orally, twice daily, morning & evening with preferably 12 hours (not less than 6 hours) between doses.
  Interventions: Drug: Tapentadol Extended Release

INTERVENTIONS:
Drug: Tapentadol Extended Release — Tablet taken orally, twice daily, morning & evening with preferably 12 hours (not less than 6 hours) between doses. Titration phase: Starting at 100 mg, increasing at a minimum of 3 day intervals by 50 mg, with a maximum dose of 250 mg.
  Other Names: Palexia; Nucynta; Yantil
  Arms: Matching Placebo after Tapentadol in Titration Phase; Tapentadol Prolonged Release
Drug: Matching Placebo after Tapentadol in the Titration Phase. — Tablet taken orally, twice daily, morning & evening with preferably 12 hours (not less than 6 hours) between doses. In the maintenance phase only to participants that were randomized to tapentadol in the titration phase.
  Arms: Matching Placebo after Tapentadol in Titration Phase
Drug: Morphine Sulphate Controlled Release — Capsule taken orally, twice daily, morning & evening with preferably 12 hours (not less than 6 hours) between doses. Titration phase: Starting at 40 mg, increasing at a minimum of 3 days intervals by 20 mg, with a maximum dose of 100 mg. Maintenance phase: continuing on dose level established in titration phase.
  Other Names: MST® CONTINUS®
  Arms: Morphine Controlled Release

SUMMARY:
The purpose of this study will be to determine whether tapentadol (CG5503) is effective and safe in the treatment of chronic tumor related pain compared to placebo. In addition tapentadol (CG5503) will also be compared to morphine controlled release, also referred to as slow release (SR).

*Tapentadol prolonged-release (PR) is the term used in the European Union and is referred to as extended release (ER) in the United States.

DETAILED DESCRIPTION:
Normally chronic tumor related pain is controlled when participants receive repeated doses of opioid analgesics. However, opioid therapy is commonly associated with side effects such as nausea, vomiting, sedation, constipation, addiction, tolerance, and respiratory depression. Tapentadol (CG5503), a newly synthesized drug with an prolonged release (PR) formulation, also acts as a centrally acting pain reliever but has 2 mechanisms of action. The aim of this trial is to investigate the effectiveness (level of pain control) and safety (side effects) of tapentadol (CG5503) PR compared with no drug (placebo) and corresponding dose of morphine (an opioid commonly used to treat tumor related pain). This trial is a randomized, double-blind (neither investigator nor patient will know which treatment was received), active- and placebo-controlled, parallel-group, randomized withdrawal design, multicenter trial.

The trial includes a 2 week titration phase starting with either 40 mg morphine (PR) bid (bid = twice daily dosing, one dose in the morning and one dose in the evening) or 100 mg tapentadol (CG5503) PR bid. Based on effectiveness and side effects subjects can up-titrate in steps of 50 mg tapentadol (CG5503 PR) to a maximal dose of 250 mg tapentadol (CG5503) PR bid or 100 mg morphine PR bid. If participants meet the stabilisation criteria at the end of the titration phase they will be re-randomized to either placebo or active treatment and will continue 4 weeks at the last dose level in the maintenance phase. Only participants on tapentadol in the titration phase will be re-randomized to either matching placebo or to tapentadol. To maintain the blinding nature of the trial participants in the morphine arm during the titration phase will also be re-randomized however they will all remain on morphine controlled release in the maintenance phase. Placebo to match tapentadol tablets, as well as placebo to match morphine capsules, will be used to mask the treatment allocation.

Participants will be issued with an electronic diary (eDiary) to capture Numeric Rating Scale (NRS) pain intensities.

Assessments of pain relief include the pain intensity numeric rating scale (NRS) and patient global impression of change (PGIC). Safety evaluations include monitoring of adverse events, physical examinations, clinical laboratory tests and electrocardiograms. Venous blood samples will be collected for the determination of serum concentrations of tapentadol (CG5503).

ELIGIBILITY:
Inclusion Criteria

* Male and non-pregnant, non-lactating female subjects.
* Of at least 18 years of age with chronic malignant tumor-related pain with a mean pain intensity (NRS) of 5 points or higher.
* Subjects who are opioid-naïve or pretreated with an equianalgesic dose range equivalent of up to 160 mg oral morphine per day and are dissatisfied with prior treatment.
* Women must be postmenopausal, surgically sterile, or practicing or agree to practice an effective method of birth control throughout the trial.
* Expected course of the disease and the pain that would permit compliance with the trial protocol over the entire trial period.

Exclusion Criteria

Key Exclusion Criteria:

* Subjects will be excluded from the study if they have a history of seizure disorder or epilepsy;
* known history and/or presence of cerebral tumor or cerebral metastases.
* history of alcohol or drug abuse;
* uncontrolled hypertension,
* clinical laboratory values reflecting severe renal insufficiency,
* moderate or severe hepatic impairment,
* hepatitis B or C, HIV,
* inadequate bone marrow reserve
* currently treated with radiotherapy,
* pain-inducing chemotherapy,
* anti-parkinsonian drugs, neuroleptics, monoamine oxidase inhibitors, serotonin norepinephrine reuptake inhibitor (SNRI) or any other analgesic therapy than investigational medication or rescue medication during the trial.
* selective serotonin reuptake inhibitor (SSRI) treatments are allowed if taken for at least 30 days before the screening period of the study at an unchanged dose.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 622 (Actual)
Dates: Start 2007-07; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hans Georg Kress, Dr., Principal Investigator — Clinic of Anaesthesiology and Pain Management, AKH Vienna
Locations (71):
- Austria (4):
  - Site 043004, Klagenfurt
  - Site 043002, Vienna
  - Site 043001, Vienna
  - Site 043005, Vienna
- Bulgaria (6):
  - Site 359013, Gabrovo
  - Site 359011, Pleven
  - Site 359014, Plovdiv
  - Site 359004, Shumen
  - Site 359008, Sofia
  - Site 359012, Varna
- Croatia (6):
  - Site 385007, Osijek
  - Site 385001, Slavonski Brod
  - Site 385004, Varaždin
  - Site 385006, Zabok
  - Site 385002, Zagreb
  - Site 385003, Zagreb
- Czechia (7):
  - Site 420005, Brno
  - Site 420002, České Budějovice
  - Site 420006, Hradec Králové
  - Site 420007, Liberec
  - Site 420008, Olomouc
  - Site 420001, Pilsen
  - Site 420004, Prague
- Site 033101, Tarbes, France
- Germany (7):
  - Site 049009, Berlin
  - Site 049012, Cologne
  - Site 049014, Essen
  - Site 049007, Löwenstein
  - Site 049020, Potsdam
  - Site 049006, Waldkirch
  - Site 049002, Wiesbaden
- Hungary (7):
  - Site 036001, Debrecen
  - Site 036005, Komárom
  - Site 036003, Mátraháza
  - Site 036002, Nyíregyháza
  - Site 036010, Szekszárd
  - Site 036006, Székesfehérvár
  - Site 036009, Székesfehérvár
- Site 039001, Napoli, Italy
- Moldova (2):
  - Site 373001, Chisinau
  - Site 373002, Chisinau
- Poland (4):
  - Site 048004, Bydgoszcz
  - Site 048005, Gdansk
  - Site 048007, Poznan
  - Site 048001, Warsaw
- Romania (7):
  - Site 040006, Brasov
  - Site 040002, Bucharest
  - Site 040003, Bucharest
  - Site 040004, Bucharest
  - Site 040005, Cluj-Napoca
  - Site 040001, Iași
  - Site 040007, Timișoara
- Russia (5):
  - Site 007010, Arkhangelsk
  - Site 007003, Moscow
  - Site 007007, Nizhny Novgorod
  - Site 007012, Vladikavkaz
  - Site 007005, Yaroslavl
- Serbia (5):
  - Site 381003, Belgrade
  - Site 381004, Belgrade
  - Site 381005, Belgrade
  - Site 381001, Kamenitz
  - Site 381002, Niš
- Slovakia (2):
  - Site 421005, Banská Bystrica
  - Site 421001, Košice
- Spain (6):
  - Site 034009, Barcelona
  - Site 034005, Barcelona
  - Site 034006, Maó
  - Site 034012, Pamplona
  - Site 034004, Seville
  - Site 034002, Valencia
- Site 046001, Stockholm, Sweden

REFERENCES:
- [Result] Kress HG, Koch ED, Kosturski H, Steup A, Karcher K, Lange B, Dogan C, Etropolski MS, Eerdekens M. Tapentadol prolonged release for managing moderate to severe, chronic malignant tumor-related pain. Pain Physician. 2014 Jul-Aug;17(4):329-43. PMID 25054392
- [Result] Kress HG, Koch ED, Kosturski H, Steup A, Karcher K, Dogan C, Etropolski M, Eerdekens M. Direct conversion from tramadol to tapentadol prolonged release for moderate to severe, chronic malignant tumour-related pain. Eur J Pain. 2016 Oct;20(9):1513-8. doi: 10.1002/ejp.875. Epub 2016 Apr 7. PMID 27062079

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial started on 13 Jun 2007 with the enrollment of the first participant and was completed on 04 Jun 2012 with the last follow-up examination. 622 participants signed informed consent. 505 participants were randomized and 504 had at least one dose of trial medication. 496 participants were part of the safety analysis set.
Pre-assignment Details: One site was excluded from all analysis sets (efficacy and safety) due to GCP non-compliance. Thus 8 participants who were randomized and treated are not reported in the tables below.
  The participants in the tapentadol titration phase were re-randomized to tapentadol or placebo in the maintenance phase.
Groups:
- Morphine Controlled Release: Oral Morphine 40 mg to 100 mg twice daily. Capsule taken orally, twice daily, morning & evening with preferably 12 hours (not less than 6 hours) between doses.
- Matching Placebo After Tapentadol in Titration Phase: Oral Tapentadol 100 mg to 250 mg twice daily. Participants randomized to placebo received 100 mg tapentadol prolonged release (PR) twice daily for 3 days to taper them off the tapentadol dose they had received in the Titration Phase. From the 4th day (Day 18) all participants received matching placebo in the maintenance (i.e. randomized withdrawal) phase.
Period: Titration Phase
Arm/Group | Tapentadol Prolonged Release | Morphine Controlled Release | Matching Placebo After Tapentadol in Titration Phase
Started | 338 | 158 | 0 (All participants in the titration phase were in the tapentadol arm during the titration phase.)
Completed | 279 | 129 | 0
Not Completed | 59 | 29 | 0
Not completed — Adverse Event | 22 | 12 | 0
Not completed — Death | 4 | 2 | 0
Not completed — Lack of Efficacy | 10 | 0 | 0
Not completed — Withdrawal by Subject | 16 | 13 | 0
Not completed — Trial Medication non-compliant | 4 | 1 | 0
Not completed — Other | 3 | 1 | 0
Period: Discontinuations After Titration Phase
Arm/Group | Tapentadol Prolonged Release | Morphine Controlled Release | Matching Placebo After Tapentadol in Titration Phase
Started | 279 | 129 | 0
Completed | 218 (Participants meeting stabilization criteria on days 13-15 in the titration phase were re-randomized.) | 109 (Participants meeting stabilization criteria on days 13-15 in the titration phase were re-randomized.) | 0
Not Completed | 61 | 20 | 0
Not completed — Adverse Event | 6 | 0 | 0
Not completed — Lack of Efficacy | 48 | 17 | 0
Not completed — Withdrawal by Subject | 2 | 2 | 0
Not completed — Trial Medication non-compliant | 0 | 1 | 0
Not completed — Other | 5 | 0 | 0
Period: Maintenance Phase
Arm/Group | Tapentadol Prolonged Release | Morphine Controlled Release | Matching Placebo After Tapentadol in Titration Phase
Started | 106 (106 of 218 participants in the tapentadol titration arm were re-randomized and treated.) | 109 | 112 (112 of 218 participants in the tapentadol titration arm were re-randomized and treated.)
Completed | 89 | 93 | 95
Not Completed | 17 | 16 | 17
Not completed — Adverse Event | 5 | 6 | 6
Not completed — Death | 3 | 0 | 2
Not completed — Lack of Efficacy | 2 | 2 | 4
Not completed — Withdrawal by Subject | 6 | 7 | 3
Not completed — Trial medication non-compliant | 0 | 0 | 1
Not completed — Resolution of pain | 0 | 0 | 1
Not completed — Other | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Titration Phase:
  Safety Analysis Set (N = 496) Full Analysis Set (N = 492)
  Maintenance Phase:
  Safety Analysis Set (N = 327) Full Analysis Set (N = 325)
  Note:
  One site was excluded from all analysis sets (efficacy and safety) due to GCP non-compliance. Thus 8 participants who were randomized and treated are not reported in the tables below.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tapentadol Prolonged Release | Morphine Controlled Release | Total
Number analyzed (Participants) | 338 | 158 | 496
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 224 | 102 | 326
  >=65 years | 114 | 56 | 170
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.8 (10.39) | 61.5 (10.21) | 60.4 (10.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 150 | 75 | 225
  Male | 188 | 83 | 271
Region of Enrollment [Number; unit: participants]
  Austria | 5 | 3 | 8
  Bulgaria | 21 | 13 | 34
  Croatia | 27 | 11 | 38
  Czech Republic | 12 | 3 | 15
  France | 1 | 0 | 1
  Germany | 33 | 14 | 47
  Hungary | 40 | 21 | 61
  Italy | 1 | 0 | 1
  Moldova, Republic of | 14 | 5 | 19
  Poland | 24 | 13 | 37
  Romania | 47 | 21 | 68
  Russian Federation | 51 | 26 | 77
  Serbia | 37 | 19 | 56
  Slovakia | 4 | 1 | 5
  Spain | 18 | 6 | 24
  Sweden | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Scored as Responder in Maintenance Phase.
Description: A "responder" is a participant in the study that:
  1. completed 28 days of the maintenance phase
  2. had a numeric rating scale score below 5 on the 11 point scale (where 0 indicates no pain and 10 indicates worst possible pain. This twice daily current pain score was averaged over Day 18 to Day 43.
  3. did not use more than 20 mg of rescue medication per day on average in the 28 day maintenance period (from Day 18 to Day 43).
  A participant that met all 3 of the above-mentioned criteria is counted as a responder, in other words the participant benefited from the assigned drug treatment. A participant that failed to meet only 1 of the 3 criteria is not counted as a responder.
Time Frame: Day 18 through Day 43 (End of Maintenance Phase)
Population: Full Analysis Set (Maintenance Phase).
Measure: Number; unit: participants
Groups:
- Tapentadol Prolonged Release (Maintenance Phase): Oral Tapentadol 100 mg to 250 mg twice daily. Tablet taken orally, twice daily, morning & evening with preferably 12 hours (not less than 6 hours) between doses. The participant continued at the dose that was effective at the end of the Titration Phase.
- Morphine Controlled Release (Maintenance Phase): Oral Morphine 40 mg to 100 mg twice daily. Capsule taken orally, twice daily, morning & evening with preferably 12 hours (not less than 6 hours) between doses. The participant continued at the dose that was effective at the end of the Titration Phase.
Arm/Group | Tapentadol Prolonged Release (Maintenance Phase) | Morphine Controlled Release (Maintenance Phase) | Matching Placebo After Tapentadol in Titration Phase
Number analyzed (Participants) | 105 | 109 | 111
participants | 65 | 75 | 55

2. Secondary Outcome: Average Daily Pain Intensity Scores, Averaged Per Week by Treatment, During the Titration Phase in the Tapentadol Treatment Arm.
Description: Participants were asked to record their "average pain over the last 24 hours" pain intensity each evening. Average pain scores are the averages of all scores recorded during each week. The participant scored their pain intensity on an 11-point Numerical Rating Scale (NRS) where a score of 0 indicated "no pain" and a score of 10 indicated "pain as bad as you can imagine".
Time Frame: Day 1 through Day 14 (End of Titration Phase)
Population: Full Analysis Set (Titration Period), observed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tapentadol Prolonged Release
Number analyzed (Participants) | 329
units on a scale
  Prior to start of the Titration Phase: number analyzed (Participants) | 282
  Prior to start of the Titration Phase | 6.315 (1.4435)
  End of Week 1 of the Titration Phase | 5.324 (1.7476)
  End of Week 2 of the Titration Phase: number analyzed (Participants) | 295
  End of Week 2 of the Titration Phase | 4.021 (1.6872)

3. Secondary Outcome: Average Daily Pain Intensity Scores, Averaged Per Week by Treatment, During the Titration Phase in the Morphine Treatment Arm.
Description: as for outcome 2
Time Frame: Day 1 through Day 14 (End of Titration Phase)
Population: Full Analysis Set (Titration Period), observed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Morphine Controlled Release
Number analyzed (Participants) | 156
units on a scale
  Prior to start of the Titration Phase: number analyzed (Participants) | 135
  Prior to start of the Titration Phase | 6.162 (1.5693)
  End of Week 1 of the Titration Phase | 4.906 (1.9039)
  End of Week 2 of the Titration Phase: number analyzed (Participants) | 135
  End of Week 2 of the Titration Phase | 3.669 (1.7851)

4. Secondary Outcome: Average Daily Pain Intensity Scores, Averaged Per Week by Treatment, During the Maintenance Phase.
Description: as for outcome 2
Time Frame: Day 18 through Day 43 (End of Maintenance Phase)
Population: Full Analysis Set (Maintenance Period). Last observation carried forward.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Matching Placebo After Tapentadol in the Titration Phase: Oral Tapentadol 100 mg to 250 mg twice daily. Participants randomized to placebo in the maintenance phase received 100 mg tapentadol prolonged release twice daily for 3 days to taper them off the tapentadol dose they had received in the Titration Phase. From the 4th day (Day 18) all participants received matching placebo in the maintenance (i.e. randomized withdrawal) phase.
- Morphine Controlled Release: Oral Morphine 40 mg to 100 mg twice daily. Capsule taken orally, twice daily, morning & evening with preferably 12 hours (not less than 6 hours) between doses. The participant continued at the dose that was effective at the end of the Titration Phase.
Arm/Group | Tapentadol Prolonged Release (Maintenance Phase) | Matching Placebo After Tapentadol in the Titration Phase | Morphine Controlled Release
Number analyzed (Participants) | 105 | 111 | 109
units on a scale
  Prior to start of Maintenance Phase | 3.198 (1.2043) | 2.928 (1.2353) | 2.928 (1.4106)
  End of Week 1 of the Maintenance Phase | 3.220 (1.2385) | 3.115 (1.3799) | 2.903 (1.4645)
  End of Week 2 of the Maintenance Phase | 3.248 (1.3724) | 3.005 (1.5723) | 2.858 (1.4783)
  End of Week 3 of the Maintenance Phase | 3.129 (1.3267) | 3.055 (1.6702) | 2.775 (1.4312)
  End of Week 4 of the Maintenance Phase | 3.121 (1.3768) | 3.095 (1.7349) | 2.768 (1.5065)

5. Secondary Outcome: Current Pain Intensity Scores, Averaged Per Week, During the Titration Phase in the Tapentadol Arm.
Description: Participants were asked to record their current pain intensity in the morning and evening. Average pain scores are the averages of all scores recorded during each week. The participant scored their pain intensity on an 11-point Numerical Rating Scale (NRS) where a score of 0 indicated "no pain" and a score of 10 indicated "pain as bad as you can imagine".
Time Frame: Day 1 through Day 14 (End of Titration Phase)
Population: Full Analysis Set (Titration Phase), observed.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Tapentadol Prolonged Release (Titration Phase): Oral Tapentadol 100 mg to 250 mg twice daily. Tablet taken orally, twice daily, morning & evening with preferably 12 hours (not less than 6 hours) between doses.
Arm/Group | Tapentadol Prolonged Release (Titration Phase)
Number analyzed (Participants) | 331
units on a scale
  Start of Titration: number analyzed (Participants) | 320
  Start of Titration | 6.344 (1.4568)
  End of Week 1 | 5.326 (1.7650)
  End of Week 2: number analyzed (Participants) | 302
  End of Week 2 | 4.049 (1.8015)

6. Secondary Outcome: Current Pain Intensity Scores, Averaged Per Week, During the Titration Phase in the Morphine Arm.
Description: Participants were asked to record their current pain intensity in the morning and evening. Average pain scores are the averages of all scores recorded during the during each week. The participant scored their pain intensity on an 11-point Numerical Rating Scale (NRS) where a score of 0 indicated "no pain" and a score of 10 indicated "pain as bad as you can imagine".
Time Frame: Day 1 through Day 14 (End of Titration Phase)
Population: Observed, i.e. participants contributing data via their electronic diary.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Morphine Controlled Release (Titration Phase): Oral Morphine 40 mg to 100 mg twice daily. Capsule taken orally, twice daily, morning & evening with preferably 12 hours (not less than 6 hours) between doses.
Arm/Group | Morphine Controlled Release (Titration Phase)
Number analyzed (Participants) | 157
units on a scale
  Start of Titration: number analyzed (Participants) | 150
  Start of Titration | 6.258 (1.5609)
  End of Week 1 | 4.937 (1.9080)
  End of Week 2: number analyzed (Participants) | 136
  End of Week 2 | 3.690 (1.8365)

7. Secondary Outcome: Current Pain Intensity Scores, Averaged Per Week by Treatment, During the Maintenance Phase.
Description: Participants were asked to record their current pain intensity in the morning and evening. Average pain scores are the averages of all scores recorded during the 3 days prior to re-randomization or during each week. The participant scored their pain intensity on an 11-point Numerical Rating Scale (NRS) where a score of 0 indicated "no pain" and a score of 10 indicated "pain as bad as you can imagine".
Time Frame: Day 15 through Day 43 (End of Maintenance Phase)
Population: Full Analysis Set (Maintenance Period). Last observation carried forward.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tapentadol Prolonged Release (Maintenance Phase) | Matching Placebo After Tapentadol in the Titration Phase | Morphine Controlled Release
Number analyzed (Participants) | 105 | 111 | 109
units on a scale
  Prior to start of maintenance phase | 3.1444 (1.16485) | 2.8686 (1.19387) | 2.832 (1.3895)
  End of Week 1 | 3.0869 (1.22550) | 3.0073 (1.32110) | 2.780 (1.3706)
  End of Week 2 | 3.1148 (1.27905) | 2.8683 (1.47838) | 2.790 (1.4170)
  End of Week 3 | 3.0137 (1.26515) | 2.9122 (1.60299) | 2.733 (1.4512)
  End of Week 4 | 3.0002 (1.37551) | 2.9220 (1.68601) | 2.728 (1.4481)

8. Secondary Outcome: Use of Rescue Medication in the Titration Phase.
Description: The number of participants using rescue medication morphine sulfate immediate release 10 mg tablets in the titration phase were counted. This data was captured in an electronic diary.
  During the trial, morphine immediate release 10 mg was allowed as required without a maximum dose defined. However, participants were only re-randomized if their mean consumption of rescue medication was less or equal to 2 doses (20 mg) per day during the last 3 days of the titration phase).
Time Frame: Day 1 through Day 14 (End of Titration Phase)
Population: Full Analysis Set (Titration phase), observed.
Measure: Number; unit: participants
Arm/Group | Tapentadol Prolonged Release | Morphine Controlled Release
Number analyzed (Participants) | 335 | 157
participants | 241 | 91

9. Secondary Outcome: Number of Participants Using Immediate Release Morphine Rescue Medication in the Maintenance Phase
Description: Participants were issued morphine 10 mg immediate release medication. The number of participants using rescue medication morphine sulfate immediate release 10 mg tablets in the maintenance phase were counted. This use of morphine immediate release was captured in each participant's electronic diary.
Time Frame: Day 15 through Day 43 (End of Maintenance Phase)
Population: Full Analysis Set (Maintenance phase), observed.
Measure: Number; unit: participants
Groups:
- Tapentadol Prolonged Release: Oral Tapentadol 100 mg to 250 mg twice daily. Tablet taken orally, twice daily, morning & evening with preferably 12 hours (not less than 6 hours) between doses. The participant continued at the dose that was effective at the end of the Titration Phase.
Arm/Group | Tapentadol Prolonged Release | Morphine Controlled Release | Matching Placebo After Tapentadol in Titration Phase
Number analyzed (Participants) | 105 | 109 | 111
participants | 75 | 67 | 80

10. Secondary Outcome: The Average Mean Total Daily Dose of Rescue Medication.
Description: Mean total daily dose of rescue medication morphine sulphate immediate release tablets in milligrams per day (mg/day).
Time Frame: Day 1 (Start of Titration Phase) through Day 43 (End of Maintenance Phase)
Population: Full analysis set for each phase of the trial, observed.
Measure: Mean (Standard Deviation); unit: milligrams per day of morphine rescue
Groups:
- Morphine Controlled Release Titration Phase: Oral Morphine 40 mg to 100 mg twice daily. Capsule taken orally, twice daily, morning & evening with preferably 12 hours (not less than 6 hours) between doses
- Matching Placebo After Tapentadol in Titration Phase: Oral Tapentadol 100 mg to 250 mg twice daily in the titration phase. Followed by matching placebo in the maintenance (i.e. randomized withdrawal phase).
- Morphine Controlled Release Maintenance Phase: Oral Morphine 40 mg to 100 mg twice daily. Capsule taken orally, twice daily, morning & evening with preferably 12 hours (not less than 6 hours) between doses. The participant continued at the dose that was effective at the end of the Titration Phase.
Arm/Group | Tapentadol Prolonged Release (Titration Phase) | Morphine Controlled Release Titration Phase | Tapentadol Prolonged Release (Maintenance Phase) | Matching Placebo After Tapentadol in Titration Phase | Morphine Controlled Release Maintenance Phase
Number analyzed (Participants) | 335 | 157 | 105 | 111 | 109
milligrams per day of morphine rescue | 13.31 (17.41) | 8.87 (12.50) | 11.2 (12.739) | 13.65 (13.666) | 8.91 (14.951)

11. Secondary Outcome: Changes in the Short Form 36® Health Survey (SF-36®) During the Titration Phase.
Description: The Short Form 36 (SF-36) includes several brief questions on 8 aspects, (physical functioning, role physical, bodily pain, general health, vitality, social functioning, role-emotional and mental health) that a participant was asked to score over the last week. Low scores on the Physical Component Summary measure indicate limitations in physical functioning, e.g. a high degree of bodily pain and physical limitations etc. For the Mental Component Summary measure, a low score is indicative of frequent psychological distress, social and role disability due to emotional problems etc. The theoretical range for the physical component score is 12.3279 to 59.6503. The theoretical range for the mental component score is 13.5313 to 59.6503. Positive values for changes in the component scores indicate an improvement.
Time Frame: Day 1 (Start of Titration); Day 14 (End of Titration Phase)
Population: Full analysis set (Titration Period), observed. Start of Titration and Endpoint Titration observations.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tapentadol Prolonged Release | Morphine Controlled Release
Number analyzed (Participants) | 285 | 131
units on a scale
  Mental Component Summary | 1.3 (10.63) | 1.1 (11.78)
  Physical Component Summary | 2.0 (5.99) | 3.1 (6.48)

12. Secondary Outcome: Changes in the Short Form 36® Health Survey (SF-36®) During the Maintenance Phase.
Description: as for outcome 11
Time Frame: Day 15 (Start of Maintenance); Day 43 (End of Maintenance Phase)
Population: Full analysis set (Maintenance Phase), observed. Start of Maintenance and Endpoint Maintenance observations.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Tapentadol Extended Release: Oral Tapentadol 100 mg to 250 mg twice daily. Tablet taken orally, twice daily, morning & evening with preferably 12 hours (not less than 6 hours) between doses. The participant continued at the dose that was effective at the end of the Titration Phase.
Arm/Group | Tapentadol Extended Release | Morphine Controlled Release | Matching Placebo After Tapentadol in Titration Phase
Number analyzed (Participants) | 95 | 97 | 103
units on a scale
  Mental Component Summary | -0.4 (10.81) | -2.164 (9.42) | -1.5 (9.99)
  Physical Component Summary | -1.1 (6.26) | -0.671 (7.21) | -0.9 (6.29)

13. Secondary Outcome: Change in the EuroQoL (EQ-5D) Health Status Index (United Kingdom Time Trade-off Value Set) Change From Start of Titration to Endpoint Titration.
Description: The participant scores the EuroQol-5D. The EuroQoL-5D is a five dimensional health state classification. Each dimension is assessed on a 3-point ordinal scale (1 = no problems, 2 = some problems, 3 = extreme problems).
  The responses to the five EQ-5D dimensions are scored using a utility-weighted algorithm to derive an EQ-5D health status index score between 0 to 1, with 1.00 indicating "full health" and 0 representing dead. A positive change in the mean indicates that during this phase the health status improved. A positive change indicates an improvement in health. The minimal important difference is 0.074 (range -0.011 to 0.140).
Time Frame: Day 1 (Start of Titration); Day 14 (End of Titration Phase)
Population: Full analysis set (Titration Phase), observed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tapentadol Prolonged Release | Morphine Controlled Release
Number analyzed (Participants) | 286 | 132
units on a scale | 0.093 (0.3294) | 0.131 (0.3162)

14. Secondary Outcome: Health Related Quality of Life: EuroQol-5D Health State Visual Analog Scale (VAS) Titration Phase.
Description: EuroQoL-5D Health State Visual Analog Scale (VAS) is a participant rated questionnaire to assess health-related quality of life in terms of a single index value. The VAS component rates current health state on a scale from 0 (worst imaginable health state) to 100 (best imaginable health state); higher scores indicate better health. The values indicated represent the change from Day 1, a positive value indicates an improvement since the start of treatment.
Time Frame: Day 1 (Start of Titration); Day 14 (End of Titration Phase)
Population: Full analysis set (Titration Phase), observed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tapentadol Prolonged Release | Morphine Controlled Release
Number analyzed (Participants) | 286 | 131
units on a scale | 3.8 (22.63) | 5.6 (20.42)

15. Secondary Outcome: Change in the EuroQoL (EQ-5D) Health Status Index (United Kingdom Time Trade-off Value Set) Over Time in the Maintenance Phase for Tapentadol and the Placebo Randomized Withdrawal Treatment Arms.
Description: The participant scores the EuroQol-5D. The EuroQoL-5D is a five dimensional health state classification. Each dimension is assessed on a 3-point ordinal scale (1 = no problems, 2 = some problems, 3 = extreme problems).
  The responses to the five EQ-5D dimensions are scored using a utility-weighted algorithm to derive an EQ-5D health status index score between 0 to 1, with 1.00 indicating "full health" and 0 representing dead. A negative change in the mean indicates a worsening in health status since the beginning of the maintenance phase. A positive change indicates an improvement in health. The minimal important difference in the Health Status Index is 0.074 (range -0.011 to 0.140).
Time Frame: Day 15 (Start of Maintenance); Day 43 (End of Maintenance Phase)
Population: Full Analysis Set (Maintenance Phase), observed. Start of Maintenance and Endpoint Maintenance observations. No morphine treatment analysis was planned.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tapentadol Prolonged Release | Matching Placebo After Tapentadol in Titration Phase
Number analyzed (Participants) | 95 | 103
units on a scale | -0.0626 (0.3130) | -0.058 (0.2909)

16. Secondary Outcome: Changes in Health Related Quality of Life: EuroQol-5D Health State Visual Analog Scale (VAS) Maintenance Phase.
Description: EuroQoL-5D Health State Visual Analog Scale (VAS) is a participant rated questionnaire to assess health-related quality of life in terms of a single index value. The VAS component rates current health state on a scale from 0 (worst imaginable health state) to 100 (best imaginable health state); higher scores indicate a better health state. The values indicated represent the change from Day 15, a negative mean value indicates a worsening of health-related quality of life since the start of the maintenance phase.
Time Frame: Day 15 (Start of Maintenance); Day 43 (End of Maintenance Phase)
Population: Full Analysis Set (Maintenance Phase), observed. Start of Maintenance and Endpoint Maintenance observations.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tapentadol Prolonged Release | Morphine Controlled Release | Matching Placebo After Tapentadol in the Titration Phase
Number analyzed (Participants) | 95 | 97 | 103
units on a scale | -2.1 (19.80) | -0.6 (16.94) | -1.5 (18.55)

17. Secondary Outcome: Patient Global Impression of Change
Description: In the Patient Global Impression of Change (PGIC) the participant is asked "Since I began study treatment, my overall status is". The participant is asked to circle one of seven categories. Scores range from very much improved to very much worse. The question was asked at the end of the maintenance phase with reference to the start of the maintenance phase where the participant continued at the dose that was effective at the end of the Titration Phase.
Time Frame: Day 43 (End of Maintenance Phase)
Population: Full Analysis Set, observed.
Measure: Number; unit: participants
Arm/Group | Tapentadol Prolonged Release | Morphine Controlled Release | Matching Placebo After Tapentadol in Titration Phase
Number analyzed (Participants) | 94 | 97 | 103
participants
  Very Much Improved | 4 | 6 | 6
  Much Improved | 29 | 23 | 31
  Minimally Improved | 33 | 38 | 38
  No Change | 10 | 12 | 11
  Minimally Worse | 10 | 6 | 9
  Much Worse | 7 | 12 | 7
  Very Much Worse | 1 | 0 | 1

18. Secondary Outcome: Quality of Sleep (Sleep Questionnaire) in the Titration Phase.
Description: Participants were asked the following question: "Please rate the overall quality of your sleep last night?" The quality of sleep from the start of the titration phase to the end of the titration phase was measured. The participant could choose one of the following options: Excellent, good, fair and poor.
Time Frame: Day 1 (Start of Titration); Day 14 (end of Titration Phase)
Population: Full Analysis Set (Titration Phase), observed. Tapentadol: 302 participants dosed gave a response at the start of titration and from 309 participants at the end of titration.
  Morphine: 143 participants dosed gave a response at the start of titration and from 142 participants at the end of titration.
Measure: Number; unit: participants
Arm/Group | Tapentadol Prolonged Release | Morphine Controlled Release
Number analyzed (Participants) | 338 | 158
participants
  Excellent at the start of the titration phase | 9 | 4
  Excellent at the end of the titration phase | 12 | 3
  Good at the start of the titration phase | 77 | 47
  Good at the end of the titration phase | 139 | 64
  Fair at the start of the titration phase | 142 | 51
  Fair at the end of the titration phase | 121 | 61
  Poor at the start of the titration phase | 74 | 41
  Poor at the end of the titration phase | 37 | 14
  Not completed at the start of titration | 36 | 15
  Not completed at the end of the titration | 29 | 16

19. Secondary Outcome: Quality of Sleep (Sleep Questionnaire) During the Maintenance Phase of the Trial.
Description: Participants were asked the following question: "Please rate the overall quality of your sleep last night?" The quality of sleep from the start of maintenance to the completion of treatment is reported. The participant could choose one of the following options: Excellent, good, fair and poor.
Time Frame: Day 15 (Start of Maintenance); Day 43 (End of Maintenance Phase)
Population: FAS (Maintenance Phase) Last Observation Carried Forward for participants re-randomized.
  Tapentadol: 105 participants responded at the start and 103 participants at the end.
  Morphine: 108 participants responded at the start and 107 participants at the end.
  Placebo: 110 participants responded at the start and 107 participants at the end.
Measure: Number; unit: participants
Arm/Group | Tapentadol Prolonged Release | Morphine Controlled Release | Matching Placebo After Tapentadol in Titration Phase
Number analyzed (Participants) | 105 | 108 | 110
participants
  Excellent at start of maintenance phase | 8 | 2 | 4
  Excellent at the end of maintenance phase | 8 | 9 | 8
  Good at start of maintenance phase | 55 | 51 | 60
  Good at the end of maintenance phase | 43 | 40 | 49
  Fair at start of maintenance phase | 35 | 50 | 42
  Fair at the end of maintenance phase | 38 | 53 | 37
  Poor at start of maintenance phase | 7 | 5 | 4
  Poor at the end of maintenance phase | 14 | 5 | 13

20. Secondary Outcome: Clinical Opioid Withdrawal Scale (COWS) at the End of the Titration Phase.
Description: This instrument was developed by the National Institute on Drug Abuse. The physical components of withdrawal are primarily evaluated and based on questions and clinical observations. The possible opioid withdrawal effects are assessed using the Clinical Opioid Withdrawal Score (COWS). The COWS is a clinician rated 11-item scale that primarily evaluates the physical components of opioid withdrawal and is based on questions and clinical observations. Responses are rated on a Likert-type scale ranging from 0 to 4 or 5 depending on the item. The total COWS score is the sum of all individual items.
  The following withdrawal categories are based on the total COWS score:
  * None: total score below 5;
  * Mild: total score from 5 to 12;
  * Moderate: total score 13 to 24;
  * Moderately Severe: total score 25 to 36;
  * Severe: total score above 36. The investigator completes the COWS after participants discontinued trial medication 2 to less than 5 days after last intake of trial medication.
Time Frame: Day 14 (End of Titration Phase)
Population: Safety Analysis Set (Titration Phase). Participants that took at least one dose of trial medication in the titration phase, and discontinued trial medication at the end or during the titration phase and did not continue on other opioid medication.
Measure: Number; unit: participants
Groups:
- Matching Placebo After Tapentadol in Titration Phase: Oral Tapentadol 100 mg to 250 mg twice daily. Followed by matching placebo in the maintenance (i.e. randomized withdrawal phase).
Arm/Group | Tapentadol Prolonged Release | Morphine Controlled Release | Matching Placebo After Tapentadol in Titration Phase
Number analyzed (Participants) | 7 | 6 | 9
participants
  None | 7 | 5 | 8
  Mild | 0 | 1 | 1
  Moderate | 0 | 0 | 0
  Moderately Severe | 0 | 0 | 0
  Severe | 0 | 0 | 0

21. Secondary Outcome: Clinical Opioid Withdrawal Score (COWS) at the End of the Maintenance Phase.
Description: as for outcome 20
Time Frame: Day 43 (End of Maintenance Phase)
Population: Safety Analysis Set. Participants that did not discontinue due to adverse event during the first week of the maintenance phase and started opioid after last study medication.
Measure: Number; unit: participants
Arm/Group | Tapentadol Prolonged Release | Morphine Controlled Release | Matching Placebo After Tapentadol in Titration Phase
Number analyzed (Participants) | 26 | 29 | 29
participants
  None | 19 | 23 | 21
  Mild | 7 | 6 | 8
  Moderate | 0 | 0 | 0
  Moderately Severe | 0 | 0 | 0
  Severe | 0 | 0 | 0

22. Secondary Outcome: Change in the Patient Assessment of Constipation Symptoms (PAC-SYM) During the Titration Phase
Description: The Constipation Assessment (PAC-SYM) is a 12-item self-report questionnaire that assesses the severity of symptoms of constipation. Participants are asked "How severe have each of these symptoms been in the last two weeks?" e.g. "Pain in your stomach". There are 3 subscales: 4 questions on Abdominal symptoms, 3 questions on rectal symptoms and 5 questions on stool symptoms. Responses are rated on a 5-point Likert Scale ranging from 0 (absence of symptom) to 4 (very severe symptoms). The changes in overall mean and in each of the mean sub-scores vary theoretically from -4 to +4 (where a change of +4 would indicate a change from not present to very severe symptom). If the changes in the overall or subscale mean scores are positive then there is a worsening in symptoms associated with constipation from the start to the end of the titration phase.
Time Frame: Day 1 (Start of Titration); Day 14 (End of Titration Phase)
Population: Per Protocol Set (Titration Phase), observed. Start of Titration and Endpoint Titration observations.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tapentadol Prolonged Release | Morphine Controlled Release
Number analyzed (Participants) | 216 | 93
units on a scale
  Overall abdominal subscale | -0.062 (0.6507) | -0.076 (0.7242)
  Overall rectal subscale | 0.059 (0.6442) | -0.006 (0.6736)
  Overall stool subscale | 0.02 (0.812) | 0.13 (0.870)
  Overall PAC-SYM score | 0.003 (0.5782) | 0.027 (0.6154)

23. Secondary Outcome: Change in the Patient Assessment of Constipation Symptoms (PAC-SYM) During the Maintenance Phase
Description: The Constipation Assessment (PAC-SYM) is a 12-item self-report questionnaire that assesses the severity of symptoms of constipation. Participants are asked "How severe have each of these symptoms been in the last two weeks?" e.g. "Pain in your stomach". There are 3 subscales: 4 questions on Abdominal symptoms, 3 questions on rectal symptoms and 5 questions on stool symptoms. Responses are rated on a 5-point Likert Scale ranging from 0 (absence of symptom) to 4 (very severe symptoms). The changes in overall mean and in each of the mean sub-scores vary theoretically from -4 to +4 (where a change of +4 would indicate a change from not present to very severe symptom). If the changes in the overall or subscale mean scores are positive then there is a worsening in symptoms associated with constipation from the start to the end of the maintenance phase. A negative mean change indicates an improvement.
Time Frame: Day 15 (Start of Maintenance); Day 43 (End of Maintenance Phase)
Population: Safety Analysis Set (Maintenance Phase), observed. Start of Maintenance and Endpoint Maintenance observations.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tapentadol Prolonged Release | Morphine Controlled Release | Matching Placebo After Tapentadol in Titration Phase
Number analyzed (Participants) | 95 | 96 | 103
units on a scale
  Overall abdominal subscale | -0.105 (0.6280) | 0.026 (0.5966) | -0.075 (0.5330)
  Overall rectal subscale | 0.017 (0.5086) | 0.014 (0.5090) | -0.033 (0.5822)
  Overall stool subscale | -0.07 (0.743) | 0.03 (0.724) | -0.03 (0.667)
  Overall PAC-SYM score | -0.059 (0.4992) | 0.024 (0.4584) | -0.048 (0.4771)

ADVERSE EVENTS:
Time Frame: Serious adverse events reported any time after treatment is taken, to within 30 days after end of treatment.
Groups:
- Tapentadol Prolonged Release (Maintenance Phase): Oral Tapentadol 100 mg to 250 mg twice daily. The participant continued at the dose that was effective at the end of the Titration Phase.
- Morphine Controlled Release (Maintenance Phase): Oral Morphine 40 mg to 100 mg twice daily. The dose that was effective at the end of the Titration Phase.
Arm/Group | Tapentadol Prolonged Release (Titration Phase) | Morphine Controlled Release (Titration Phase) | Tapentadol Prolonged Release (Maintenance Phase) | Matching Placebo After Tapentadol in Titration Phase | Morphine Controlled Release (Maintenance Phase)
Serious Adverse Events (participants affected / at risk) | 25/338 | 6/158 | 12/106 | 10/112 | 6/109
Other Adverse Events (participants affected / at risk) | 112/338 | 80/158 | 41/106 | 34/112 | 37/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tapentadol Prolonged Release (Titration Phase) (N=338) | Morphine Controlled Release (Titration Phase) (N=158) | Tapentadol Prolonged Release (Maintenance Phase) (N=106) | Matching Placebo After Tapentadol in Titration Phase (N=112) | Morphine Controlled Release (Maintenance Phase) (N=109)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 1 | 4 | 2 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Trismus (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 0
Hospitalization due to travel problems (General disorders) | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Cor pulmonale acute (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Superior vena cava syndrome (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 1
Adrenocortical insufficiency acute (Endocrine disorders) | 1 | 0 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Female genital tract fistula (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Death (General disorders) | 0 | 0 | 2 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 1 | 0 | 0
Cardiovascular insufficiency (Cardiac disorders) | 0 | 0 | 2 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Blood urea increased (Investigations) | 0 | 0 | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Lobar pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Withdrawal syndrome (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tapentadol Prolonged Release (Titration Phase) (N=338) | Morphine Controlled Release (Titration Phase) (N=158) | Tapentadol Prolonged Release (Maintenance Phase) (N=106) | Matching Placebo After Tapentadol in Titration Phase (N=112) | Morphine Controlled Release (Maintenance Phase) (N=109)
Nausea (Gastrointestinal disorders) | 42 | 38 | 16 | 17 | 11
Constipation (Gastrointestinal disorders) | 48 | 28 | 12 | 13 | 12
Vomiting (Gastrointestinal disorders) | 17 | 25 | 8 | 3 | 6
Dry Mouth (Gastrointestinal disorders) | 4 | 10 | 3 | 2 | 1
Dizziness (Nervous system disorders) | 17 | 10 | 5 | 4 | 0
Somnolence (Nervous system disorders) | 14 | 10 | 3 | 2 | 6
Fatigue (General disorders) | 10 | 8 | 4 | 6 | 6
Decreased Appetite (Metabolism and nutrition disorders) | 9 | 6 | 8 | 6 | 6
Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 6 | 2 | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 9 | 7 | 4 | 1 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor reserves the right to review any publication pertaining to the trial at least 30 days before it is submitted for publication. Neither party has the right to prohibit publication unless publication can be shown to affect possible patent rights.